CLINICAL TRIAL: NCT04198155
Title: Renal Denervation Using Stereotactic Radiotherapy System for the Treatment of Refractory Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19XHCR20D
Record Dates: First submitted 2019-12-11; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- stereotactic body radiotherapy (SBRT) (Experimental): Noninvasive SBRT will be delivered in a single fraction to bilateral renal arteries determined by CT-guidance.
  Interventions: Radiation: stereotactic body radiotherapy (SBRT)

INTERVENTIONS:
Radiation: stereotactic body radiotherapy (SBRT) — Image-guided stereotactic body radiation therapy

SUMMARY:
This study is conducted to investigate the short-term safety and preliminary efficacy of stereotactic radiotherapy for renal denervation to treat refractory hypertension.

DETAILED DESCRIPTION:
This will be a single centre, single arm, prospective cohort study. Patients with refractory hypertension will receive single fraction stereotactic radiotherapy for renal denervation. The study has been designed in a careful and stepwise dose escalation fashion in order to minimize the potential risks associated with this innovative technique. The dose escalation is guided by 3+3 algorithm to ensure more patients will be spared dose limiting toxicities and more patients will be entered on the dose level that will be chosen as optimal dose of maximal effect. Low dosing levels with established safety profile will first be applied before administering higher dosing levels based on preclinical studies.

Safety is the primary endpoint of this study. Safety will be assessed by incidence and evaluation of any serious adverse events using CTCAE v5.0 criteria associated with the procedure through 90 days. Efficacy will be evaluated by assessing mean reduction in average 24-hour ambulatory blood pressure at 90 days post-treatment.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 55 and ≤ 75 years. Systolic blood pressure of 160 mmHg or greater despite being treated with at least three hypertensive drugs for more than 3 months.

Exclusion Criteria:

GFR < 45 ml/min/1.73 m2. Known causes of secondary hypertension. Hospitalized for hypertensive crisis within 1 year. History of acute coronary syndrome or cerebrovascular accident within the last 6 months.

Pregnancy or have a pregnancy plan. Contrast media or iodine allergy. History of abdominal radiotherapy or adhesive intestinal obstruction. Severe valvular heart disease. Stenosis >50% or renal artery aneurysm in either renal artery. Others.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | 90 days
  Safety will be assessed by incidence and evaluation of any serious adverse events using CTCAE v5.0 criteria that are related to the procedure.
Ambulatory Blood Pressure Reduction | 90 days
  Mean reduction in average 24-hour ambulatory blood pressure at 90 days post-treatment

SECONDARY OUTCOMES:
Office Blood Pressure Reduction | 90 days
  Mean reduction in office blood pressure at 90 days post-treatment
Number of Drug Adjustments | 90 days
  Number of drug adjustments for hypertension through 90 days after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Gang Li, MD, Principal Investigator — Xinhua Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Xinhua Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No